CLINICAL TRIAL: NCT01161758
Title: A Crossover Study on the Effect of Cervical Mobilization on Motor Function and Pressure Pain Threshold in Pain Free Individuals
Brief Title: Study on the Effect of Cervical Mobilization on Motor Function and Pressure Pain Threshold in Pain Free Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Curtin University (Other)
Responsible Party: Prof Anthony Wright, Curtin University of Technology
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: PT0004
Record Dates: First submitted 2010-07-08; First posted 2010-07-14 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2005-11

CONDITIONS: Neck Pain
Keywords: physical therapy; pain threshold; electromyography; musculoskeletal manipulation; neck muscles
MeSH Terms: conditions — Neck Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Passive cervical mobilisation (Active Comparator): Grade III cervical mobilization technique as described by Maitland. Applied to left C5/6 Segment.
  Interventions: Other: Passive cervical mobilisation
- Manual contact (Placebo Comparator): Manual contact control, which involved light manual contact on the left C5/C6 segment as if to perform the treatment technique.
  Interventions: Other: Manual contact
- Non-contact control (No Intervention): Non-contact control, which involved the subject resting in the treatment position without any physical contact between the researcher and the subject.

INTERVENTIONS:
Other: Passive cervical mobilisation — Passive cervical mobilization which involved an oscillatory grade III unilateral postero-anterior mobilization applied to the left C5/C6 segment. The mobilization consisted of 3 periods of 1 minute applications with a resting period of 1 minute in between.
  Other Names: Physiotherapy
  Arms: Passive cervical mobilisation
Other: Manual contact — Manual contact control, which involved light manual contact on the left C5/C6 segment as if to perform the treatment technique. The light manual contact consisted of 3 periods of 1 minute applications with a resting period of 1 minute in between.
  Other Names: placebo light touch
  Arms: Manual contact

SUMMARY:
Passive accessory cervical mobilization is widely used as a clinical approach to the management of musculoskeletal pain of spinal origin. The purpose of the study is to determine if passive cervical mobilization can improve motor function in situations where motor performance is not impaired by the presence of pain.

DETAILED DESCRIPTION:
Cervical mobilization has been shown to elicit effects on pain perception, autonomic function and motor function in subjects who experience musculoskeletal pain. The improvement in motor function may be a direct effect of the treatment or secondary to a hypoalgesic effect. This study aims to demonstrate whether it is possible to alter motor function following joint mobilization, in situations where motor performance is not impaired by pain.

ELIGIBILITY:
Inclusion Criteria:

* No history of neck or back pain over the last six months
* Without any previous experience with spinal manual therapy techniques

Exclusion Criteria:

* History of musculoskeletal or rheumatologic conditions
* Any kind of spinal surgery
* Dizziness
* Previous trauma to the cervical spine
* Neurological signs or symptoms

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-04; Primary Completion 2005-10 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Electromyography of sternocleidomastoid muscle. | Pre intervention (baseline) and 1 minute post intervention
  Measurement of sternocleidomastoid muscle activation during deep neck flexion. The degree of neck flexion is determined by a pressure biofeedback unit place underneath the neck. EMG of the left and right sternocleidomastoids are recorded for 5seconds at each level of neck flexion

SECONDARY OUTCOMES:
Pressure pain threshold | Pre intervention (baseline) and 1 minute post intervention
  The algometer to measure pressure pain threshold was applied at a constant rate of 40 kPa/sec on the posterior aspect of the left and right articular pillar of C5/C6.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Soon Tze Chin, MManipTher, Principal Investigator — The University of Queensland; Annina Schmid, MManipTher, Principal Investigator — The University of Queensland; Elias Fridriksson, MManipTher, Principal Investigator — Curtin University; Philip Cheong, MManipTher, Principal Investigator — Curtin University; Elisabeth Gresslos, MManipTher, Principal Investigator — Curitn University of Technology; Anthony Wright, PhD, Study Chair — Curtin University